CLINICAL TRIAL: NCT01466257
Title: Detection of DNA Mutations in Head and Neck Squamous Cell Carcinoma
Brief Title: Biomarkers in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000715520; ECOG-E5397T2
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IVA squamous cell carcinoma of the larynx; stage IVA squamous cell carcinoma of the lip and oral cavity; stage IVA squamous cell carcinoma of the oropharynx; stage IVA squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVB squamous cell carcinoma of the larynx; stage IVB squamous cell carcinoma of the lip and oral cavity; stage IVB squamous cell carcinoma of the oropharynx; stage IVB squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVC squamous cell carcinoma of the larynx; stage IVC squamous cell carcinoma of the lip and oral cavity; stage IVC squamous cell carcinoma of the oropharynx; stage IVC squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: DNA analysis of tumor tissue may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the mutation rates of HRAS and PIK3CA in patients with head and neck squamous cell carcinoma (HNSCC) who were treated with cisplatin/placebo and cisplatin/cetuximab on protocol ECOG-E5397.
* To determine the association between HRAS or PIK3CA mutation status and clinical benefits (i.e., response, progression-free survival, and overall survival) in patients treated with cisplatin/cetuximab compared with those receiving cisplatin/placebo on protocol ECOG-E5397.

OUTLINE: DNA is isolated from one unstained slide per patient. The mutations in HRAS and PIK3CA are determined using BEAMING technology.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Treated on protocol ECOG-E5397

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E5397
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
Mutation rates of HRAS and PIK3CA | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Christine H. Chung, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins